CLINICAL TRIAL: NCT04342468
Title: Relationship of Blood Pressure Variability and Cardiovascular Disease Events Among Patients With Hypertension
Brief Title: Blood Pressure Variability and Cardiovascular Disease Events in Patients With Hypertension
Acronym: BPV
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Professor Chia Yook Chin, Professor, University of Malaya
Other Study IDs: 2017314-5047; WI207736 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Blood Pressure Variability; Hypertension; Cardiovascular Diseases
Keywords: blood pressure variability; Hypertension; cardiovascular diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-interventional — No intervention

SUMMARY:
Cardiovascular Disease (CV) including stroke is the leading cause of death in Malaysia Hypertension is a major contributor to this. Prevalence of hypertension in Malaysia is high (42%) in adults age 30 years or older. Besides the actual blood pressure (BP) level recently, blood pressure variability (BPV) has been recognized as an independent and strong predictor of CV events especially strokes. However, data on the BP variability and its relationship to CV events is very limited in Asia, particularly in Malaysia. Hence the investigators aim to study BPV and its relationship to CV events in treated hypertensive patients

DETAILED DESCRIPTION:
This will be a cross-sectional study on patients with hypertension. The 10-year retrospective data on BP, treatment, biochemical changes, kidney function and CV events will be extracted from patient records.

Eligible patients who have given written informed consent will be given a questionnaire capturing data of their socio-demographic status, weight, height and BP measured.

Those agreeable to measure their own BP at home 3 times a day for a week will be loaned a BP device to measure their own BP at home. The home BP readings will be recorded onto a provided form and returned to the investigators.

Data will be analysed to

1. determine BPV of the clinic visit-to-visit BPV (long tem BPV)
2. determine the day to day BPV (short term BPV)
3. examine the BPV to CV events, kidney function, cognition
4. determine the prevalence of white coat and masked hypertension
5. determine the level of control of BP
6. examine the relationship of ownership of home BP devices to control and satisfaction of treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients on treatment for hypertension of at least 3 years
* Patients who consent to the study

Exclusion Criteria:

* those unable to give consent
* recent (less than 6 months) of cardiovascular events (stroke, heart attack, heart failure)
* patients on dialysis
* patients with end stage kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with hypertension on follow up at the primary care clinic of University of Malaya Medical Centre who fulfill the inclusion and exclusion criteria are eligible to be enrolled into the study
  Eligible patients were recruited in a consecutive manner
Sampling Method: Non-Probability Sample
Enrollment: 1736 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The standard deviation value of blood pressure variability in treated hypertensive patients | 31 Dec 2020
  The various indices of day-to-day and long term Blood pressure variability will be calculated giving the actual BPV (in absolute number ) in these patients
Percentage of cardiovascular events in those with higher BPV compared to those with lower BPV | 31 Dec 2020
  BPV will be categorized as above or below the mean BPV of the entire group. The number of CV events in percentage in each group will be compared It is expected that those with higher BPV will have more CV events

SECONDARY OUTCOMES:
Percentage of Treated hypertensives with White Coat or Masked hypertension | 31 Dec 2020
  The Home and Clinic BP measurements will be used to determine the percentage of Masked and White Coat Hypertension. These two conditions are expected to be associated with more CV events than those with control of both clinic and home BP.
Difference in cognition in those with higher BP variability compared to those with lower BPV | 31 Dec 2020
  The Montreal Cognitive Assessment (MoCA) score will be compared between those with higher with those with lower BPV. The minimum MoCA score is 0 and the maximum is 30. A higher MoCA score indicates better cognition. A MoCA score of 26 is considered as normal. The MoCA score is expected to be lower in those with higher BPV.

CONTACTS AND LOCATIONS:
Overall Officials: Lai M Looi, MBBS FRCPath, Study Director — University of Malaya Medical Centre
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
The data are only useful for this study

REFERENCES:
- [Background] Mancia G. Short- and long-term blood pressure variability: present and future. Hypertension. 2012 Aug;60(2):512-7. doi: 10.1161/HYPERTENSIONAHA.112.194340. Epub 2012 Jun 25. No abstract available. PMID 22733459
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Sever PS, Poulter NR. Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. Lancet. 2010 Mar 13;375(9718):895-905. doi: 10.1016/S0140-6736(10)60308-X. PMID 20226988
- [Background] Muntner P, Joyce C, Levitan EB, Holt E, Shimbo D, Webber LS, Oparil S, Re R, Krousel-Wood M. Reproducibility of visit-to-visit variability of blood pressure measured as part of routine clinical care. J Hypertens. 2011 Dec;29(12):2332-8. doi: 10.1097/HJH.0b013e32834cf213. PMID 22025235
- [Background] Rogers MA, Small D, Buchan DA, Butch CA, Stewart CM, Krenzer BE, Husovsky HL. Home monitoring service improves mean arterial pressure in patients with essential hypertension. A randomized, controlled trial. Ann Intern Med. 2001 Jun 5;134(11):1024-32. doi: 10.7326/0003-4819-134-11-200106050-00008. PMID 11388815
- [Background] Chia YC, Ching SM, Lim HM. Visit-to-visit SBP variability and cardiovascular disease in a multiethnic primary care setting: 10-year retrospective cohort study. J Hypertens. 2017 May;35 Suppl 1:S50-S56. doi: 10.1097/HJH.0000000000001333. PMID 28350621
- [Background] Chia YC, Lim HM, Ching SM. Long-Term Visit-to-Visit Blood Pressure Variability and Renal Function Decline in Patients With Hypertension Over 15 Years. J Am Heart Assoc. 2016 Nov 7;5(11):e003825. doi: 10.1161/JAHA.116.003825. PMID 27821404